CLINICAL TRIAL: NCT02912858
Title: Intermittent Pneumatic Compression of the Foot vs Geko Plus R-2 Neuromuscular Electrostimulation Device in Venous Leg Ulcer Patients: Comparison of Effects on Lower Limb Circulation
Brief Title: Intermittent Pneumatic Compression of the Foot vs Geko Plus R-2 Neuromuscular Electrostimulation Device in Venous Leg Ulcer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study withdrawn
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FKD-IPC-003
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- geko plus R-2 (Experimental): neuromuscular electrostimulation
  Interventions: Device: geko plus R-2

INTERVENTIONS:
Device: geko plus R-2 — The gekoTM plus R-2 devices (acting on the common peroneal nerve) and IPC devices will be activated for 10mins prior to measuring blood flow.
  The sequence of application of IPC and gekoTM plus R-2 devices will be randomly selected with 10 minutes recovery between active therapies.

SUMMARY:
Chronic venous leg ulcers (VLU) are painful, debilitating wounds that place a significant burden on the patient, their family, and healthcare resources. Treating VLU can present a significant challenge to clinicians, who currently have a limited range of treatments at their disposal. The mainstay of treatment is compression bandaging, ambulation and elevation at rest. In addition to the aforementioned, intermittent pneumatic compression has also been utilised1. When applied to the leg or foot intermittent pneumatic compression (IPC) devices intermittently inflate and deflate to increase venous return. These devices can be uncomfortable to wear, and compliance can be inhibited because of size, weight and external power source that limit the patient's mobility. In patients who cannot walk, or in those who are unable to tolerate compression bandaging, ulcers may deteriorate and never heal. Accordingly, there is a need for novel, alternative devices or strategies that can be used to complement or replace compression bandage therapy.

DETAILED DESCRIPTION:
This is a single-centre randomised intra-patient comparison of gekoTM plus R-2 R-2 and IPC.

Blood flow will be measured after each device has been activated for 10 minutes with a 10 minute rest between devices to allow blood flow to return to baseline. The order the devices will be fitted is determined randomly. Activation of the device for 10 minutes before measurement is deemed appropriate as previous studies have demonstrated significant increases in blood flow following as little as five minutes use of the devices.

In this short study the standard of care (typically compression bandaging), will be suspended temporarily to allow the fitting of the gekoTM plus R-2 and IPC devices in order to measure blood flow. This is not seen as a risk to the patient as the device is only in operation for 30 minutes plus 10 minutes rest within the care pathway.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Intact healthy skin at the site of device application
3. Able to understand the Patient Information Sheet
4. Willing and able to give informed consent
5. Willing and able to follow the requirements of the protocol
6. Subjects who had a chronic venous leg ulcer (i.e. CEAP classification of C6 1) greater than 2 cm2 and less than 10 cm in maximum diameter,
7. ABPI of 0.8-1.2 inclusive

Exclusion Criteria:

1. Wound infection either acute or chronic
2. History of significant haematological disorders or DVT with the preceding six months
3. Pregnant
4. Pacemakers or implantable defibrillators
5. Use of any other neuro-modulation device
6. Current use of TENS in pelvic region, back or legs
7. Use of investigational drug or device within the past 4 weeks that may interfere with this study
8. Recent surgery that may affect the study (such as abdominopelvic, or lower limb) in the opinion of the investigator.
9. Recent trauma to the lower limbs
10. Size of leg incompatible with the gekoTM plus R-2 device
11. Obesity (BMI > 34)
12. Any medication deemed to be significant by the Investigator
13. Subjects who had an index venous leg ulcer greater in maximum diameter than 10cm in any one dimension, or less than 2cm.
14. Diabetes
15. Clinical evidence of peripheral arterial disease (i.e signs or symptoms, in the opinion of the researcher)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The lower limb blood flow between gekoTM plus R-2 and IPC devices in VLU patients will be assessed. | 3 months
  Duplex ultrasound of the femoral vein and artery will be performed with bilateral recording of blood flow velocity. After 10 minutes activation of either geko™ or IPC and after the 10 minutes the devices will swapped over and measurements performed. All measurements to be carried out in triplicate.

SECONDARY OUTCOMES:
Adverse events assessments | 3 months
  Patients will be monitored for adverse events throughout the duration of the study. Adverse events may be spontaneously reported by the subject, observed by the study personnel.
  Serious Adverse Events will be reported to the Sponsor, the National Research Ethics Service (NRES) recognised Research Ethics Committee.

IPD SHARING:
Plan to Share IPD: Yes